CLINICAL TRIAL: NCT04109963
Title: Trial of Remote Ischemic Pre-Conditioning in Vascular Cognitive Impairment
Acronym: TRIC-VCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Consortium on Neurodegeneration in Aging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB19-0861
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-08

CONDITIONS: Vascular Dementia; Cerebral Small Vessel Diseases; Cerebral Small Vessel Ischaemic Disease; Vascular Cognitive Impairment
Keywords: vascular cognitive impairment, cerebral small vessel diseases, remote ischemic conditioning
MeSH Terms: conditions — Dementia, Vascular; Cerebral Small Vessel Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel arm, open-label, blinded end-point (PROBE) design.
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed masked to treatment assignment. Participants will be aware of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC once per day (Active Comparator): RIC performed once a day on one arm. Each RIC session will consist of 4 cycles of unilateral or simultaneous bilateral upper arm ischemia for 5 minutes followed by reperfusion for another 5 minutes. The procedure will be performed by using an electric auto-control device with cuffs that inflate to a pressure of 200 mmHg during the ischemic period.
  Interventions: Device: Remote ischemic conditioning
- RIC twice per day (Active Comparator): RIC performed twice a day on one arm, approximately 12 hours apart. Each RIC session will consist of 4 cycles of unilateral or simultaneous bilateral upper arm ischemia for 5 minutes followed by reperfusion for another 5 minutes. The procedure will be performed by using an electric auto-control device with cuffs that inflate to a pressure of 200 mmHg during the ischemic period.
  Interventions: Device: Remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — Remote ischemic conditioning therapy to the upper arm will be delivered by an automated device (RIC VCI) manufactured by Seagull Aps (Denmark).

SUMMARY:
Cerebral small vessel disease is a common cause of cognitive impairment. Remote ischemic pre-conditioning (RIC) is a technique to induce brief periods of limb ischemia-reperfusion that is hypothesized to increase tolerance of the brain to hypoperfusion and increase cerebral blood flow. Patients with cognitive impairment, preserved basic activities of daily living, and brain computed tomography (CT) or magnetic resonance imaging (MRI) evidence of confluent white matter hyperintensities or multiple brain infarcts will be randomized to either RIC performed once a day on one arm, or twice per day on one arm, for 30 days, to test tolerability and effects on MRI markers of blood flow.

DETAILED DESCRIPTION:
Cerebral small vessel disease (cSVD) accounts for 20-25% of all strokes and is the most common cause of vascular cognitive impairment (VCI) as well as a major contributor to mixed dementia, potentially interacting with Alzheimer's disease. Remote ischemic pre-conditioning (RIC) is a technique to induce brief periods of limb ischemia-reperfusion that is hypothesized to increase tolerance of the brain to hypoperfusion. This is a prospective, open-label randomized controlled clinical trial with blinded endpoint assessment (PROBE). Participants that complete a 14-day run-in period will be randomized to 30 days of either: a) RIC performed once per day on one arm, or b) RIC performed twice per day on one arm. Each RIC session will consist of 4 cycles of unilateral upper arm ischemia for 5 minutes followed by reperfusion for another 5 minutes, administered by modified blood pressure monitor (under an Investigational Trail Authorization from Health Canada). The primary outcome is tolerability, defined as the proportion in each trial arm that complete 80% or more of the assigned RIC sessions. Secondary outcomes will include pain scores, cognition, and MRI markers of cerebral blood flow and white matter integrity.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of cerebral small vessel disease on CT or MRI, defined as either beginning confluent white matter hypodensities/hyperintensities (ARWMC scale) or two or more supratentorial infarcts
* Montreal Cognitive Assessment <25
* Concern on the part of the patient, caregiver, or clinician that there has been a decline from previous level of cognitive functioning
* Independent with basic activities of daily living (response (a) to questions 2, 4, 5, 6, 7, 8, 9, and 14 on the Bristol Activities of Daily Living scale).

Exclusion Criteria:

* Cortical infarcts larger than 10 mm axial diameter
* Neuroimaging evidence of mass lesion, intracerebral hemorrhage, vascular malformation, or evidence of non-vascular disease such as hydrocephalus.
* Residence in long-term care facility.
* Other significant neurological or psychiatric disease (e.g. multiple sclerosis).
* Does not have a study partner who can provide corroborative information.
* English or French is not sufficiently proficient for clinical assessment and neuropsychological testing
* Montreal Cognitive Assessment score <13
* Unable to undergo MRI due to medical contraindications or inability to tolerate the procedure.
* Co-morbid medical illness that in the judgment of the study investigator makes it unlikely that the participant will be able to complete three months of study follow-up.
* On therapeutic anticoagulation with doses used for treatment of deep venous thrombosis, pulmonary embolism, or for stroke prevention in atrial fibrillation.
* Significant bleeding diathesis.
* Any symptomatic or previously known arm soft-tissue disease, vascular injury, or peripheral vascular disease
* Hypertension with systolic blood pressure >=180 mmHg despite medical treatment at the time of enrolment.
* Planned revascularization (any angioplasty or vascular surgery) within the next 3 months.
* Planned surgical procedure within the next 3 months.
* Currently receiving an investigational drug or device by other studies
* Blood pressure cuff cannot be sized properly (arm circumference is <23 cm or >42 cm)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Adherence | 30 days
  Proportion completing 80% or more sessions.

SECONDARY OUTCOMES:
Discontinuation | 30 days
  Cessation of device use
Randomization | 14 days
  Proportion completing the run-in period and proceeding to randomization
Physical examination | 30 days
  Proportion with signs of arm soft tissue or neurovascular injury
Arm deep venous thrombosis | 30 days
  Arm deep venous thrombosis
Pain | 30 days
  Mean peak and end-cycle pain levels reported using the Numeric Rating Scale for pain (based on subjective report, ranging from 0 [no pain] to 10 [worst possible pain]).
MRI cerebral blood flow | 30 days and 90 days
  Change in cerebral blood flow measured by arterial spin label MRI
MRI white matter hyperintensity volume | 30 days and 90 days
  Change in white matter hyperintensity volume on FLAIR
MRI diffusion tensor imaging | 30 days and 90 days
  Change in MRI peak skeletonized mean diffusivity
Global cognition | 30 days and 90 days
  Change in Montreal Cognitive Assessment
Neuropsychological tests | 30 days and 90 days
  Change in Trail-Making A and B
Neuropsychiatric symptoms | 30 days and 90 days
  Change in Mild Behavioural Impairment Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Eric Smith, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The completely de-identified study dataset will be posted to the University of Calgary section of the PRISM dataverse at the time of publication of the main study results in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study dataset will be made publicly available at the time of publication of the main study results in a peer-reviewed journal.
Access Criteria: Open to the public.
URL: https://dataverse.scholarsportal.info/dataverse/calgary

REFERENCES:
- [Derived] Ganesh A, Barber P, Black SE, Corbett D, Field TS, Frayne R, Hachinski V, Ismail Z, Mai LM, McCreary CR, Sahlas D, Sharma M, Swartz RH, Smith EE. Trial of remote ischaemic preconditioning in vascular cognitive impairment (TRIC-VCI): protocol. BMJ Open. 2020 Oct 14;10(10):e040466. doi: 10.1136/bmjopen-2020-040466. PMID 33055122
- Available data/document: Individual Participant Data Set: Not yet available — https://dataverse.scholarsportal.info/dataverse/calgary — The dataset with individual de-identified participant data will be hosted on the University of Calgary PRISM dataverse once the main results results are published. The identifier will be assigned when the dataset is uploaded.